CLINICAL TRIAL: NCT02634281
Title: Extended (6-Week) Varenicline Preloading: Does it Facilitate Smoking Reduction and Cessation?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0239-15-SZMC
Record Dates: First submitted 2015-12-01; First posted 2015-12-18 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Experimental): Subjects in Group A will receive varenicline for six weeks .During this phase, subjects will be asked to reduce cigarette smoking by 50 percent. At week 6 all participants will be instructed to stop smoking before receiving 12 weeks of varenicline treatment
  Interventions: Drug: Varenicline
- group B (Active Comparator): group B will receive placebo for 5 weeks and varenicline for 1 week. During this phase, subjects will be asked to reduce cigarette smoking by 50 percent. At week 6 all participants will be instructed to stop smoking before receiving 12 weeks of varenicline treatment
  Interventions: Drug: Varenicline; Drug: placebo

INTERVENTIONS:
Drug: Varenicline — Subjects in Group A will receive varenicline for six weeks while those in group B will receive placebo for 5 weeks and varenicline for 1 week. During this phase, subjects in both groups will be asked to reduce cigarette smoking by 50 percent. At week 6 all participants will be instructed to stop smoking before receiving 12 weeks of varenicline treatment
  Other Names: champix; chantix
Drug: placebo — Subjects in Group A will receive varenicline for six weeks while those in group B will receive placebo for 5 weeks and varenicline for 1 week. During this phase, subjects in both groups will be asked to reduce cigarette smoking by 50 percent. At week 6 all participants will be instructed to stop smoking before receiving 12 weeks of varenicline treatment
  Arms: group B

SUMMARY:
SUMMARY Rationale: Worldwide, cigarette smoking carries a high mortality. Since the available cessation programs are not effective for all smokers, new strategies are necessary for tobacco control.

Primary objective: To investigate whether a 6-week varenicline preloading facilitates smoking reduction and cessation compared with the standard varenicline treatment schedule.

Design: Parallel group, double-blind, randomised controlled clinical trial. Participants: Smokers of both sexes from the general population. Methods: Participants will be randomized into two groups of treatment. Subjects in Group A will receive varenicline for six weeks while those in group B will receive placebo for 5 weeks and varenicline for 1 week. During this phase, subjects in both groups will be asked to reduce cigarette smoking by 50 percent. At week 6 all participants will be instructed to stop smoking before receiving 12 weeks of varenicline treatment. Visits will be arranged at randomization, week 4, week 6 (Quit day (QD)) and at week 1, 6, 12, and 24 after QD.

Measurements: These will include vital signs, smoking history, spirometry, expired CO, salivary cotinine, nicotine dependence, and withdrawal symptoms. Primary outcome is continuous abstinence at 6 months.

Sample size: For an estimated difference of quit rates of 15% at 24 weeks (30% for group A vs. 15% for group B) 121 subjects per group are needed (Total = 242 subjects).

Statistical analysis: T tests (rational variables) and x2 test or Fisher's exact test (nominal variables) will be used as appropriate.

Expected benefits: This study might contribute to optimize the current use of varenicline.

DETAILED DESCRIPTION:
Study design:

The study is a parallel group, double-blind, randomised controlled clinical trial. Allocation to treatment will be made when the subject has been entered into the study that is when he/she has fulfilled the inclusion/exclusion criteria (see below). Visits will be arranged at inclusion, at week 4 and 6 (Quit day (QD)) after inclusion, and at week 1, 6, 12, and 24 after QD.

Study population:

Participants will be eligible smokers from throughout Jerusalem, who want to reduce then stop smoking.

Randomisation procedure:

Subjects will be computer-randomised either to an extended varenicline preload treatment or to a regular varenicline schedule. Both groups will receive an identical treatment thereafter.

Blinding:

Due to the nature of the intervention, blinding is possible only during the varenicline preload phase. During this phase, both the study team members and the participants will be blinded to treatment allocation. After week 6 all participants will be receiving the same, active treatment.

Study intervention:

After enrolment the subjects will be randomized to receive either varenicline preloading for 6 weeks (1 mg/day at week 1; 2 mg/day from week 2-6) (Group A) or placebo for 5 weeks and varenicline for 1 week (Group B). Then, subjects in both groups will receive regular treatment with varenicline for 12 weeks according to a schedule depicted on Table 2. Only minimal levels of advice and support will be given. However, all subjects will receive individualized verbal instructions regarding the general conduct of the study and the proper use of the study medication. All participants will be asked to reduce smoking by 50 percent during 6 weeks after inclusion then stop smoking altogether.

At baseline the following data will be collected:

1. Demographic assessment (age, sex, height and weight). Subjects will be weighed during all scheduled visits on the same scale throughout the study: prior to weighing, subjects will remove shoes and excess clothes.
2. Medical history
3. Physical examination
4. Vital signs (pulse, blood-pressure) will be assessed in the standard manner.
5. Spirometry: This will be carried out at baseline and end-study using an electronic spirometer and techniques currently performed at the Pulmonary Institute, Shaare Zedek Medical Center.
6. Smoking history and other smoking related information using the modified Cigarette Evaluation Questionnaire (mCEQ) .
7. Nicotine dependence evaluation using the Fagerström Test for Nicotine Dependence (FTND) .
8. CO in expired air. Expired carbon monoxide levels will be measured with a Bedfont monitor and recorded at each scheduled study visit. The subjects will be instructed to inhale deeply, do a 15 second breath hold, and produce a full, slow forced expiration through the disposable mouthpiece of the inflow valve of the monitor. Readings will be recorded in parts per million (ppm) of CO (non smokers = < 8 ppm ; smokers = > 10 to 75 ppm) .
9. Withdrawal symptoms: Will be measured using the Mood Symptoms Physical Scale (MPPS) (See Appendix) .
10. Salive Cotinine determinations: This will be carried out at 3 visits namely baseline visit, week 6 and end-trial.
11. Concomitant medication: Information about currently used medication will be collected

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years
* Currently smoking 10 cigarettes per day or more
* Having smoked 5 py or more
* Presenting a CO level in expired air ≥ 10 ppm
* Personally motivated to reduce or stop smoking and indicating a willingness to follow through with protocol requirements
* Willing to sign a statement of informed consent

Exclusion Criteria:

* Myocardial infarction within the last 3 months
* Unstable angina
* Severe cardiac arrhythmia
* Pregnancy or breast feeding
* Use of any form of smokeless tobacco or nicotine substitution
* Having followed any smoking cessation programme during the last 3 months
* Alcohol or other drug addiction
* Use of any form of smokeless tobacco or nicotine substitution
* Participation in any clinical trial within the past 3 months
* Women in childbearing age not willing to use contraception until week 12 after QD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence | from week 7 until week 24
  defined as avoidance of tobacco (not a single puff) since the quit date. It will be assessed by self-reported complete abstinence and expired CO < 10 ppm from week 7 until endpoint. The occurrence of occasional lapses after week 7 will be categorised as a failure in the main evaluation, but will not necessitate withdrawal if the subject is willing to continue and is considered by the investigators as competent to succeed.

SECONDARY OUTCOMES:
smoking reduction | from week 7 until week 24
  This will be measured by daily self-reported cigarettes per day and expired CO measures (at every visit). An efficient reduction will be defined by a diminution of at least 50% of the number of cigarettes smoked, together with a reduction in CO levels compared to baseline
Decline in pulmonary function | from week 7 until week 24
  The rate of decline of spirometric parameters will be calculated separately for quitters, continuing smokers and reducers from the two groups, pooled together.
adverse events | from week 7 until week 24
  The subjects will be asked about adverse events at each visit during treatment by an open-ended question. Serious adverse events are defined as events that are fatal or life threatening, permanently disabling, requiring or prolonging hospitalisation, cancer, congenital abnormality or overdose
Symptoms and physical signs associated with withdrawal: MPSS questionnaire | from week 7 until week 24
  MPSS questionnaire
Use of cigarettes | from week 7 until week 24
  For participants smoking at any time point the number of cigarettes smoked per day and the satisfaction (mCEQ questionnaire) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham BOHADANA, MD, Principal Investigator — Shaare zedek medical center, pulmonary institute
Locations (1):
- Shaare Zedek Medical center, Jerusalem, Israel

REFERENCES:
- [Derived] Bohadana A, Freier-Dror Y, Peles V, Babai P, Izbicki G. Extending varenicline preloading to 6 weeks facilitates smoking cessation: A single-site, randomised controlled trial. EClinicalMedicine. 2020 Feb 3;19:100228. doi: 10.1016/j.eclinm.2019.11.021. eCollection 2020 Feb. PMID 32055787